CLINICAL TRIAL: NCT00219622
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled, Six Week Study Of The Efficacy And Safety Of Tofimilast Dry Powder For Inhalation In Adults Diagnosed With Chronic Obstructive Pulmonary Disease
Brief Title: A Phase 2 Study of the Safety and Efficacy of a Tofimilast in Adult Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2641022
Record Dates: First submitted 2005-09-11; First posted 2005-09-22 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tofimilast

INTERVENTIONS:
Drug: tofimilast

SUMMARY:
This an initial proof of concept, phase to study to assess the safety and efficacy of tofimilast for the chronic maintenance treatment of adults with Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion Criteria:

* Moderate-severe COPD (GOLD 2003 definition)
* Smoking history of at least 10 pack-years

Exclusion Criteria:

* Any significant co-morbid disease, particularly cardiovascular
* Use of any maintenance therapy except short acting bronchodilators

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in FEV1 compared to placebo

SECONDARY OUTCOMES:
Change from baseline in other lung function parameters, dyspnea, quality of life compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (21):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Riverdale, Georgia
  - Pfizer Investigational Site, Stockbridge, Georgia
  - Pfizer Investigational Site, Normal, Illinois
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Lake Oswego, Oregon
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Bellingham, Washington
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Tukwila, Washington
- Argentina (4):
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Vicente López, Buenos Aires
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Buenos Aires
- Brazil (2):
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
- Chile (4):
  - Pfizer Investigational Site, Providencia, Santiago Metropolitan
  - Pfizer Investigational Site, Recoleta, Santiago Metropolitan
  - Pfizer Investigational Site, Santiago
  - Pfizer Investigational Site, ValparaÃ-so
- Pfizer Investigational Site, San José, Provincia de San José, Costa Rica
- Mexico (3):
  - Pfizer Investigational Site, MÃ©xico, D.f.
  - Pfizer Investigational Site, Monterrey, Nuevo LeÃ³n
  - Pfizer Investigational Site, Monterrey, Nuevo León

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2641022&StudyName=A+Phase+2+Study+of+the+Safety+and+Efficacy+of+a+Tofimilast+in+Adult+Patients+with+Chronic+Obstructive+Pulmonary+Disease